CLINICAL TRIAL: NCT06015217
Title: An Open-label Study to Assess Efficacy and Safety of a Healing Ointment When Used on Infants With Mild-to-moderate Diaper Rash
Brief Title: A Clinical Study to Assess the Efficacy and Safety of a Healing Ointment on Diaper Rash
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.US.SL.027
Record Dates: First submitted 2023-08-14; First posted 2023-08-29 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-08

CONDITIONS: Diaper Rash
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Intervention Model Description: This study only has a single group, and all subjects receive the same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): All subjects have mild to moderate diaper dermatitis and are given "Cetaphil Healing Ointment" to use with every diaper change.
  Interventions: Drug: "Cetaphil Healing Ointment"

INTERVENTIONS:
Drug: "Cetaphil Healing Ointment" — Subjects will use "Cetaphil Healing Ointment" on the diaper rash area with every diaper change

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety of a Healing Ointment in infants 2-24 months with mild to moderate diaper rash. The main question it aims to answer is:

• does a Healing Ointment improve skin texture and smoothness in infants with mild to moderate diaper dermatitis? Participants will use a Healing Ointment on the diaper area with every diaper change, have the Investigator perform efficacy and tolerability assessments, and complete questionnaires regarding subject satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must meet all the following criteria to be eligible for the study:

  1. Infant subjects aged 2 months to 24 months
  2. Females and males
  3. All Fitzpatrick skin types I-VI
  4. All races and ethnicities
  5. Subject diagnosed with mild-to-moderate diaper rash
  6. Subject with healthy immune systems
  7. Willing to be photographed at each visit (optional)
  8. Willing to abstain from use of any other topical diaper rash treatments (ointments, moisturizers, emollients, creams, and wipes) other than the assigned test product and skincare products that have been routinely used on the diaper area during the duration of the study
  9. Willing to continue using regular brands of face/body cleanser and not to begin use of any new skincare products other than the test product for the duration of the study
  10. Parent/legal guardian/legal guardians must be at least 18 years old and are willing and able to present proof of legal guardianship
  11. Parent/legal guardian/legal guardian with ability to read, understand and give consent for participation in the study
  12. Parent/legal guardians/legal guardians willing to sign a photography release form
  13. Parent/legal guardian/guardian must agree to adhere to the procedures and requirements of the study and to report to the site on the day(s) and at the time(s) scheduled for the assessments

Exclusion Criteria:

* The presence of any of the following exclusion criteria excluded a subject from enrollment in the study:

  1. Subject diagnosed with severe diaper rash
  2. History of allergy or hypersensitivity to any ingredient of the test product
  3. Presence of any disease or lesions near or on the area to be treated, e.g.,

     1. Inflammation, active, or chronic infection in or near the treatment area
     2. Psoriasis, eczema, rosacea, atopic dermatitis, herpes zoster/herpes simplex, and acanthosis
     3. Scars or deformities
  4. History of coexisting bacterial infections or medical conditions with uncontrolled gastrointestinal diseases and/or bowel movements
  5. History of severe elastosis and/or excessive sun exposure that, in the opinion of the Investigator, could have affected the outcome of the study
  6. Planning on having surgeries and/or invasive medical procedures during the course of the study
  7. Treatment with chemotherapy, immunosuppressive agents, inhaled corticosteroids, immunomodulatory therapy (e.g., monoclonal antibodies or antiviral treatment for human immunodeficiency virus or hepatitis C)
  8. Current use of topical corticosteroids, topical prescription, or oral antibiotics in the treatment area, or use within last 2 weeks
  9. Current use of over-the counter topical medications for diaper rash
  10. History of cancer or previous radiation near or on the treatment area
  11. Human immunodeficiency virus positive or active hepatitis
  12. Presence of dermal markings on or near the treatment area that, in the opinion of the Investigator, will interfere with the clinical assessments
  13. Any medical condition that, in the opinion of the Investigator, would make the subject unsuitable for inclusion (e.g., a chronic or relapsing, disease that may interfere with the outcome of the study)
  14. Other condition preventing the subject from entering the study in the Investigator's opinion, (e.g., subjects failing baseline assessments, subjects not likely to avoid other cosmetic treatments in the treatment area, subjects anticipated to be unavailable or incapable of understanding the study assessments or having unrealistic expectations of the treatment result).
  15. Study site personnel, close relatives of the study site personnel (e.g., parent/legal guardians, children, siblings, or spouse), or employees and close relatives of employees at the Sponsor company.
  16. Participation in any interventional clinical study within 30 days of screening

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Product Efficacy | Week 1, Week 3
  Product efficacy will be measured by Investigator's evaluation of skin's tactile smoothness, visual skin texture, and diaper dermatitis. Skin smoothness (tactile) and skin texture will be measured on a 10-point modified Griffith's scale, where 0 is the best possible condition and 9 is the worst possible condition, and diaper dermatitis will be measured on a 5-point scale, where 0 is the best possible condition and 4 is the worst possible condition. A decrease in scores indicates an improvement.

SECONDARY OUTCOMES:
Subject Satisfaction | Day 1, Week 1, Week 3
  To evaluate subject satisfaction using a Self-Assessment Questionnaire. Questionnaires will be tabulated; and the frequency and percentage of all response options will be reported for each question and time point. For questionnaire inquiries without baseline response data, a binomial (sign) test will be performed to test if the proportion of the combined designated favorable responses is equal to the combined designated unfavorable responses for each applicable question. A higher percentage of favorable responses with a significant p value indicates positive subject perceptions of the study treatment.
Product Tolerability | Week 1, Week 3
  Product tolerability will be measured by Investigator's evaluation of dryness, peeling, and edema on a 4-point analog scale, with half-point scores used as necessary to better describe the clinical condition, where 0 indicates parameter is not present and 3 indicates parameter is severe. A decrease in scores or lack of significant increase indicates tolerability/safety of the treatment product.

CONTACTS AND LOCATIONS:
Overall Officials: Latanya Benjamin, Principal Investigator — Young Skin
Locations (1):
- Young Skin MD, Coral Springs, Florida, United States

IPD SHARING:
Plan to Share IPD: No